CLINICAL TRIAL: NCT04398537
Title: The Role of Pre-deployment Retraction in Decreasing Biopsy Clip Migration During Stereotactic Breast Biopsies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Stefanie A. Woodard, Assistant Program Director, Diagnostic Radiology Residency Program Assistant Professor, Breast Imaging Section, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: R20-040
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Breast Biopsy
Keywords: stereostatic procedure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 5mm retraction of clip deployment apparatus (Experimental): The participants in this group will have clip placement 5mm in front of the biopsy site site.
  Interventions: Device: 5mm retraction of clip deployment apparatus.
- no retraction of clip deployment apparatus (Active Comparator): These participants will the clip delivered at the biopsy site.
  Interventions: Device: No retraction of clip deployment apparatus.

INTERVENTIONS:
Device: 5mm retraction of clip deployment apparatus. — Advancing the clip to the biopsy site and retracting 5 mm and then deploying. This is one method of standard of care and involves depositing the clip after retraction of the deployment apparatus 5 mm.
  Arms: 5mm retraction of clip deployment apparatus
Device: No retraction of clip deployment apparatus. — This is one method of standard of care and the clip will be deployed at the biopsy site.
  Arms: no retraction of clip deployment apparatus

SUMMARY:
This will be a single-center prospective randomized control trial that is Institutional Review Board (IRB) approved. The study plans to enroll 250 female patients presenting to the University of Alabama at Birmingham (UAB) for stereotactic biopsy. This study is a prospective and will target approximately 250 patients. This will be a HIPPA-compliant randomized control trial planned on spanning approximately six months' time. Patients will be entered into the study only based on their already scheduled stereotactic biopsy procedure. Patients will be informed of the study and they will be offered the opportunity to participate or not participate in the study. Their participation is completely voluntary. This study will not involve any intervention that is not already a part of standard care. Patients will be randomized to two groups, one group that will undergo clip placement with approximately with a 5 mm retraction of the biopsy clip post-placement and one that will involve no retraction prior to deployment.

ELIGIBILITY:
Inclusion Criteria:

- Females 18-99 of age with recommendation for stereotactic biopsy.

Exclusion Criteria:

* Non-female patients
* Patients < 18 years old
* Women who are pregnant

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2023-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Woodard, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
To be determined.

REFERENCES:
- [Derived] Eltoum N, Zamora K, Murray A, West J Jr, Willis J, Chieh A, Li Y, Li M, Park JM, Woodard S. The Role of Predeployment Retraction in Biopsy Marker Migration During Stereotactic Breast Biopsies: A Randomized Controlled Trial. J Breast Imaging. 2024 Nov 5;6(6):610-620. doi: 10.1093/jbi/wbae050. PMID 39236047

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 5mm Retraction of Clip Deployment Apparatus | no Retraction of Clip Deployment Apparatus
Started | 112 | 133
Completed | 102 | 118
Not Completed | 10 | 15
Not completed — Physician Decision | 10 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5mm Retraction of Clip Deployment Apparatus | no Retraction of Clip Deployment Apparatus | Total
Number analyzed (Participants) | 102 | 117 | 219
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 71 | 131
  >=65 years | 42 | 46 | 88
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 117 | 219
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White Non-Hispanic | 49 | 59 | 108
  White Hispanic | 0 | 1 | 1
  White Ethnicity Not reported | 3 | 2 | 5
  White Ethnicity Unknown | 0 | 2 | 2
  Black Non-Hispanic | 33 | 33 | 66
  Black Ethnicity Not Reported | 1 | 1 | 2
  Asian Non-Hispanic | 7 | 10 | 17
  Asian Ethnicity Unknown | 1 | 0 | 1
  Hispanic | 1 | 0 | 1
  Hispanic Non-Hispanic | 0 | 1 | 1
  Decline Race Non-Hispanic | 4 | 6 | 10
  Decline Race Ethnicity Not Reported | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Breast Biopsy Patients Whose Clip Migrated Greater Than 10mm From the Biopsy Site.
Description: This number of participants will be counted if their clip migrated more than 10mm from the biopsy site.
Time Frame: baseline through 1 hour (post biopsy mammogram/procedure)
Measure: Count of Participants; unit: Participants
Arm/Group | 5mm Retraction of Clip Deployment Apparatus | no Retraction of Clip Deployment Apparatus
Number analyzed (Participants) | 104 | 119
Participants | 46 | 44

2. Primary Outcome: Percentage of Breast Biopsy Patients Whose Clip Migrated Greater Than 10mm From the Biopsy Site.
Time Frame: baseline through 1 hour (post biopsy mammogram/procedure)
Measure: Count of Participants; unit: Participants
Arm/Group | 5mm Retraction of Clip Deployment Apparatus | no Retraction of Clip Deployment Apparatus
Number analyzed (Participants) | 104 | 119
Participants | 46 | 44

3. Primary Outcome: Average Distance of Clip Migration for the Arm That Received 5mm Retraction.
Time Frame: baseline through 1 hour (post biopsy mammogram/procedure)
Population: This was only measured on the 5mm retraction group
Measure: Mean (Standard Deviation); unit: mm
Groups:
- 5mm Retraction of Clip Deployment Apparatus: The participants in this group will have clip placement with retraction 5mm from biopsy site.
  5mm retraction of clip deployment apparatus.: Advancing the clip to the biopsy site and retracting 5 mm and then deploying. This is one method of standard of care and involves depositing the clip after retraction of the deployment apparatus 5 mm.
Arm/Group | 5mm Retraction of Clip Deployment Apparatus | no Retraction of Clip Deployment Apparatus
Number analyzed (Participants) | 46 | 0
mm | 12.1 (14.9) |

4. Primary Outcome: Average Distance of Clip Migration for the Arm That Did Not Receive Clip Retraction.
Time Frame: baseline through 1 hour (post biopsy mammogram/procedure)
Population: This was only measured on the control group
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 5mm Retraction of Clip Deployment Apparatus | no Retraction of Clip Deployment Apparatus
Number analyzed (Participants) | 0 | 44
mm |  | 9.8 (14.9)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | 5mm Retraction of Clip Deployment Apparatus | no Retraction of Clip Deployment Apparatus
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/117
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/117
Other Adverse Events (participants affected / at risk) | 0/102 | 0/117

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-04-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT04398537/Prot_SAP_ICF_000.pdf